CLINICAL TRIAL: NCT02364791
Title: A Phase II Prospective, Single Blinded, Randomized Trial of Hemopatch Compared to Standard Techniques to Achieve Air Leak Control After Complex Thoracic Surgical Procedures on High Risk Population for Prolonged Air Leak (> 5 Days - PAL).
Brief Title: A Phase II Prospective, Single Blinded, Randomized Trial of Hemopatch Compared to Standard Techniques to Achieve Air Leak Control After Complex Thoracic Surgical Procedures
Acronym: Hemopatch
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute, Naples (Other)
Collaborators: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other); Istituto Clinico Humanitas (Other); European Institute of Oncology (Other); Regina Elena Cancer Institute (Other); Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hemopatch
Record Dates: First submitted 2015-02-10; First posted 2015-02-18 (Estimated); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Thoracic Surgery Lung; Post-operative Thoracic Air Leak
Keywords: pulmonary resection; chest tube; segmentectomy; lobectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard treatment (Active Comparator): standard techniques to achieve air leak control after complex thoracic surgical procedures
  Interventions: Device: standard techniques used to achieve air leak control
- standard treatment plus hemopatch (Experimental): the addition of hemopatch to standard techniques to achieve air leak control after complex thoracic surgical procedures
  Interventions: Device: standard techniques used to achieve air leak control; Device: Hemopatch

INTERVENTIONS:
Device: standard techniques used to achieve air leak control
Device: Hemopatch
  Other Names: sealing hemostat
  Arms: standard treatment plus hemopatch

SUMMARY:
The purpose of this study is to explore whether the addition of Hemopatch to standard care can reduce prolonged air leaks and shorten the use of air drainage tube after surgery in thoracic lung surgery patients at high risk for prolonged air leaks.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* High risk of prolonged air leak due to at least one of the following reasons:

  * Preoperative FEV1<80%
  * DLco < 80%
  * LVRS (lung volume reduction surgery o pneumoplastica riduttiva)
  * Anticipation of intraoperative adhesions (ie, redo surgery)
  * Previous induction chemotherapy for locally advanced NSCLC
  * Chronic steroid use
  * Pleural mesothelioma
* Candidate to one of the following major thoracic surgical intervention:

  * Decortication
  * Reintervention on the same side of the previous intervention
  * Segmentectomy
  * Lobectomy with incomplete fissures on CT scan
* Written informed consent.

Exclusion Criteria:

* Pregnancy or breast-feeding
* Evidence of confusion or disorientation, or history of major psychiatric illness that may impair the patient's understanding of the Informed Consent Form or their ability to comply with study requirements
* Any unstable systemic disease (including active infections, any significant hepatic, renal or cardiovascular disease), metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates or prevents or the execution of surgery
* Known hypersensitivity to bovine proteins or brilliant blue (FD&C Blue No.1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-02; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
number of days from time of extubation to time of drainage tube removal | up to 7 days

SECONDARY OUTCOMES:
number of days to end of air leak | up to 7 days
  air leak measure are recorded every 6 hours
worst grade toxicity per patient | up to 6 weeks
  according to Common Terminology Criteria for Adverse Events version 4.0
change in quality of life | baseline, one week, one month
number of days from surgical intervention to patient discharge | up to 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Rocco, MD, FRCSEd, Principal Investigator — National Cancer Institute, Naples; Francesco Perrone, MD, PhD, Principal Investigator — National Cancer Institute, Naples
Locations (1):
- Istituto Nazionale Tumori - Fondazione "G.Pascale", IRCCS, Napoli, Italy